CLINICAL TRIAL: NCT05702580
Title: Pleural Fluid Agitation For Improving The Microbiologic Diagnostic Yield In Pleural Infection - A Comparative Feasibility Study
Brief Title: Fluid Agitation Microbiologic Yield In Pleural Infection Feasibility Study
Acronym: FLAG-PINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Salama Sadaka, Doctor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0107486
Record Dates: First submitted 2022-12-23; First posted 2023-01-27 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pleural Infection

STUDY DESIGN:
Intervention Model Description: All participants will undergo both thoracentesis techniques; the standard and the experimental pre-aspiration agitated fluid techniques
Masking Description: Laboratory personnel responsible for the microbiological and biochemical analysis will be blinded to the identity of the paired samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard thoracentesis followed by pre-aspiration fluid agitation (Experimental): Participants will undergo the standard thoracentesis followed by the experimental pre-aspiration fluid agitation technique
  Interventions: Procedure: Agitated Pleural Fluid Thoracentesis

INTERVENTIONS:
Procedure: Agitated Pleural Fluid Thoracentesis — Using a 16-18 gauge cannula, a standard thoracentesis will be performed then a sample of pleural fluid will be aspirated and rapidly flushed into the pleural space and redrawn again for a few cycles before a sample is finally drawn into the collection syringe

SUMMARY:
The goal of this study is to compare the microbiologic diagnostic yield of pre-aspiration agitated pleural fluid versus that of conventionally aspirated fluid in pleural infection patients. The main question it aims to answer is, whether fluid agitation helps to increase the microbiological yield.

DETAILED DESCRIPTION:
In pleural infection, It is suggested that the bacteria being diagnostically targeted, might more likely be residing on the pleural surface with a better blood supply and nutrition rather than being planktonic in the acidic, glucose deficient pleural fluid. The investigators thus hypothesize that an agitation of the pleural fluid prior to sample aspiration would aid in achieving a better cellular representation of the pleural space. This could have the effect of washing bacterial cells off the pleural surface as well as moving sedimented cells in the aspirated sample. This study aims to investigate whether an increase in the microbiological yield for infected pleural fluid could be achieved by a pre-aspiration agitation of the pleural fluid which would have a positive effect on management and eventual patient outcomes. Adult participants with pleural infection will undergo thoracentesis via both the standard and agitated fluid techniques guided by thoracic ultrasound. Microbiological yields will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Pleural infection based on clinical presentation, imaging or laboratory investigations and pleural fluid examination showing glucose < 40 mg/dL or pH <7.2 with lower respiratory infection or pus on aspiration
3. At least a moderate amount of pleural fluid collection (2 or more intercostal spaces on thoracic ultrasound)

Exclusion Criteria:

1. Minimal - mild pleural fluid deemed unsuitable for aspiration and agitation
2. Hemodynamic instability
3. Uncorrected coagulopathy
4. Transudative or exudative lymphocytic pleural effusion on biochemical analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of the microbiologic analysis | results within 1 week of sampling
  Percentage of samples with a positive microbiologic result among both aspiration techniques

SECONDARY OUTCOMES:
LDH level difference between both aspiration methods | results within 1 day of sampling
  Difference in LDH levels in the aspirated fluid via both techniques
Glucose level difference between both aspiration methods | results within 1 day of sampling
  Difference in glucose levels in the aspirated fluid via both techniques
Protein level difference between both aspiration methods | results within 1 day of sampling
  Difference in protein levels in the aspirated fluid via both techniques
Neutrophilic count difference between both aspiration methods | results within 1 day of sampling
  Difference in neutrophilic count in the aspirated fluid via both techniques
Lymphocytic count difference between both aspiration methods | results within 1 day of sampling
  Difference in lymphocytic count in the aspirated fluid via both techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Diseases Department, Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadaka A, Said R, Ashmawy H, Okasha H, Gharraf H. Pleural fluid agitation for improving the microbiologic diagnostic yield in pleural infection: a feasibility study. Respir Res. 2025 Apr 18;26(1):154. doi: 10.1186/s12931-025-03208-7. PMID 40251602